CLINICAL TRIAL: NCT00880880
Title: Improving the Assessment of Women's Health Through the Use of a Computerized Pelvic Floor Questionnaire
Brief Title: Improving Women's Health by Using an Electronic Pelvic Floor Questionnaire
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Sigma Xi Society (Unknown); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HS17028; 1R36HS017028-01A1 (AHRQ)
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2009-04

CONDITIONS: Urinary Incontinence; Fecal Incontinence; Pelvic Floor Disorders
Keywords: urinary incontinence; fecal incontinence; communication
MeSH Terms: conditions — Urinary Incontinence; Fecal Incontinence; Pelvic Floor Disorders; Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pre-visit e-PAQ-PF (Experimental): Participants assigned to fill out the e-PAQ-PF prior to their clinic visit. Participants will arrive early to clinic appointment and fill out e-PAQ-PF. Results will be given to clinician and participant. After their visit they will complete the post visit questionnaire.
  Interventions: Other: e-PAQ-PF
- post-visit e-PAQ-PF (No Intervention): Participants assigned to complete the e-PAQ-PF after their clinic visit. Pre-visit participants will sign consent form - but otherwise will receive no study interventions. Post-visit they will fill out e-PAQ-PF and post visit questionnaire.

INTERVENTIONS:
Other: e-PAQ-PF — Participants will fill out the e-PAQ-PF prior to their clinic visit. The e-PAQ-PF has 4 dimensions (urinary, bowel, vaginal, sexual) and asks about symptoms severity, bother of symptoms, and impact on quality of life. A copy of the results will be given to their clinician and the participant.
  Other Names: electronic personal assessment questionnaire - pelvic floor; electronic pelvic floor questionnaire
  Arms: pre-visit e-PAQ-PF

SUMMARY:
The overall goal of this study is to test whether an electronic pelvic floor questionnaire (e-PAQ-PF) will increase discussion rates of incontinence in a primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Woman
* Aged 40 and older
* Scheduled for a well visit at the Women's Health Internal Medicine West Clinic

Exclusion Criteria:

* Unable to speak English
* Unable to fill out questionnaire
* Excluded by patient's clinician prior to recruitment

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 284 (Actual)
Dates: Start 2007-08; Primary Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Mention of urinary incontinence in the clinic visit note

SECONDARY OUTCOMES:
Mention of fecal incontinence in the clinic visit note
Participant report of urinary discussion | same day (within one week of appointment)
Participant report of fecal incontinence discussion | same day (within one week of appointment)
MD/NP initiated urinary incontinence discussion (per participant report)
MD/NP initiate discussion of Fecal incontinence per participant report
Urinary Incontinence History Score (Assessed from Clinic Note)
Fecal Incontinence History Score (Assessed from Clinic Note)
Urinary Incontinence Assessment and Treatment Score (from Clinic Note)
Fecal Incontinence Assessment & Treatment Score (from Clinic Note)
Any Urinary Incontinence Treatment or Referral (per clinic note)
Any treatment or referral for fecal incontinence? (per clinic note)
Diagnostic code given - Urinary incontinence
Diagnostic code given - fecal incontinence
Urinary incontinence detected | clinic visit
fecal incontinence detected | clinic visit

CONTACTS AND LOCATIONS:
Overall Officials: Chris M Schussler-Fiorenza, MD, Principal Investigator — University of Wisconsin School of Medicine & Public Health; Ronald E Gangnon, PhD, Study Chair — University of Wisconsin, Madison; Arnold Wald, MD, Principal Investigator — University of Wisconsin School of Medicine & Public Health
Locations (1):
- UW Health Women's Health Internal Medicine West, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Schussler-Fiorenza Rose SM, Gangnon RE, Chewning B, Wald A. Increasing Discussion Rates of Incontinence in Primary Care: A Randomized Controlled Trial. J Womens Health (Larchmt). 2015 Nov;24(11):940-9. doi: 10.1089/jwh.2015.5230. PMID 26555779